CLINICAL TRIAL: NCT01753336
Title: A Phase IIIb, Prospective, Multicentre, Open-Label Extension Study To Assess Long Term Safety And Effectiveness Of Dysport® Using 2 mL Dilution In Adults With Cervical Dystonia
Brief Title: Long Term Safety And Effectiveness Of Dysport® In Adults With Cervical Dystonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-TL-52120-170
Record Dates: First submitted 2012-12-17; First posted 2012-12-20 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dysport® (Experimental): Dysport®, up to 500 units (U)/vial using 2mL dilution
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Dysport® (intramuscular injection), Up to 500 units (U)/vial using 2mL dilution, 3 treatment cycles
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of the protocol is to assess the long term safety of repeat treatment cycles of Dysport® 500 U using 2 mL dilution scheme for the treatment of Cervical Dystonia. This is an extension study to study A-TL-52120-169 (hereafter referred to as Study 169).

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in Study 169 that have no ongoing adverse events, which in the opinion of the Investigator are related to study treatment and that precludes them from receiving continuing therapy
* Completed Study 169, or completed all study visits up to and including Week 4 and in the event of an early withdrawal after Week 4 have ≤15% reduction in TWSTRS total score at Week 4 compared to their baseline TWSTRS total score in the double-blind study, and in the Investigator's clinical judgment, would benefit from Dysport® for CD

Exclusion Criteria:

* Diagnosis of pure retrocollis or pure anterocollis
* Requirement for Botulinum Neurotoxin (BoNT) injection to site(s) for disorders other than CD and unable to avoid such treatment(s) for the duration of the study
* Known hypersensitivity to BoNT or related compounds, or any component in the study drug formulation
* Allergy to cow's milk protein
* Myasthenia gravis, other disease of the neuromuscular junction or clinically significant, persistent neuromuscular weakness, or disease or symptoms that could interfere with the TWSTRS scoring
* Total body weight <95 lbs (43.09 kg)
* Previous phenol injections to the neck muscles
* Previous myotomy or denervation surgery involving the neck or shoulder region or deep brain stimulation to treat CD
* Cervical contracture that limited passive range of motion
* Physiotherapy initiated <4 weeks before study entry or expected to be initiated during the study
* Treatment with aminoglycoside antibiotics within 30 days prior to study treatment
* Current or expected requirement for concomitant medication that could interfere with the evaluation of study treatment
* Pregnant and/or lactating females
* Females of childbearing potential with a positive prestudy urine pregnancy test (a positive urine pregnancy test could be confirmed by a serum pregnancy test at the discretion of the investigator) and subjects, or their partners, who did not agree to use adequate contraception (hormonal or barrier method of birth control) prior to injection of study treatment and for the duration of study participation. Nonchildbearing potential is defined as postmenopause for at least 1 year, surgical sterilisation at least 3 months before entering the study, or hysterectomy
* Individuals who had family or employee relationship to study site staff or sponsor staff involved in the conduct of the study
* Any medical condition that could, as judged by the investigator, compromise compliance with the objectives and procedures of this protocol or preclude the administration of BoNT, including swallowing and other respiratory abnormality.
* Subjects who were unable and/or unwilling to comply fully with the protocol and the study instructions, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2013-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Neurology, M.D., Study Director — Ipsen
Locations (41):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Movement Disorders Center of Arizona, LLC, Scottsdale, Arizona
  - University of Arizona, Tucson, Arizona
  - East Bay Physician's Group, Berkeley, California
  - Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Loma Linda University Healthcare, Department of Neurology, Loma Linda, California
  - USC Keck School of Medicine, Los Angeles, California
  - Sutter Cancer Center, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - Advanced Neurosciences Research, Fort Collins, Colorado
  - Associated Neurologist of Southern CT, PC, Fairfield, Connecticut
  - Yale Medical Group, Yale University, New Haven, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida
  - Emerald Coast Center for Neurological Disorders, Pensacola, Florida
  - Parkinson's Treatment Center of SW Florida, Port Charlotte, Florida
  - USF HealthParkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Guilford Neurologic Associates, West Palm Beach, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Kansas City Bone & Joint Clinic, Kansas City, Kansas
  - International Clinical Research Institute, Overland Park, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Rehabilitation Consultants, PA, Eagan, Minnesota
  - University of Medicine and Dentistry of New Jersey, Stratford, New Jersey
  - Atlantic Neuroscience Institute, Summit, New Jersey
  - Kingston Neurological Associates, Kingston, New York
  - The Ichan School of Medicine at Mount Sinai, New York, New York
  - Island Neurological Associates, Plainview, New York
  - Guilford Neurologic Associates; Cone Health Medical Group, Greensboro, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati Physicians Company, LLC, Cincinnati, Ohio
  - OHSU Center for Health and Healing, Portland, Oregon
  - Penn State Hershey Neurology, Hershey, Pennsylvania
  - Coastal Neurology, PA, Port Royal, South Carolina
  - North Texas Movement Disorders Institute, Bedford, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Puget Sound Neurology, Tacoma, Washington

REFERENCES:
- [Derived] Dashtipour K, Wietek S, Rubin B, Maisonobe P, Bahroo L, Trosch R. AbobotulinumtoxinA using 2-mL dilution (500 U/2-mL) maintains durable improvement across multiple treatment cycles. J Clin Mov Disord. 2020 Aug 31;7:8. doi: 10.1186/s40734-020-00090-x. eCollection 2020. PMID 32884828
- See also: A-TL-52120-169 — https://clinicaltrials.gov/ct2/show/NCT01753310?term=A-TL-52120-169&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open label extension (OLE) study for study A-TL-52120-169 (Study 169). First subject enrolled: 14 March 2013; last subject completed: 13 October 2015. A-TL-52120-170 (Study 170) was conducted in 36 centres in the United States that had participated in Study 169 and enrolled adult subjects with cervical dystonia (CD).
Pre-assignment Details: Subjects who completed Study 169 and had no on-going Adverse Events (AEs) or whose Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) total score between Weeks 4 and 8 was reduced by ≤15% from baseline were invited to participate in this OLE study. 112 of the 134 subjects in Study 169 were enrolled into Study 170 (signed informed consent).
Groups:
- Total Dysport®: Subjects received up to 3 doses of Dysport® 500 Units (U)/vial, 2 millilitre (mL) dilution on Day 1 of up to 3 treatment cycles. Subjects who were botulinum neurotoxin (BoNT) treatment naïve at the start of Study 169 received a starting dose of 500 U/2 mL Dysport®, and subjects who were non-naïve to BoNT treatment received the same dose they had received on Day 1 of Study 169. Subjects received Dysport® by intramuscular injection into the same neck muscles that had been used for injection in Study 169. Retreatment occurred every 12 to 16 weeks, dependent on the investigator's clinical judgment. Follow-up visits occurred at Weeks 4 and 12 of each treatment cycle. Subjects were determined to have completed the study at Week 12 of Treatment Cycle 3. Dysport® contains the neurotoxin Clostridium botulinum toxin type A haemagglutinin complex (abobotulinumtoxinA).
Period: Overall Study
Arm/Group | Total Dysport®
Started | 112
Cycle 1 | 112
Cycle 2 | 98
Cycle 3 | 93
Completed | 92
Not Completed | 20
Not completed — Patient decision | 12
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 2
Not completed — Sponsor's decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all subjects who received at least 1 dose of study treatment, regardless of the amount of study treatment administered, and who had at least 1 safety record post-treatment or attended a post-treatment visit.
Groups:
- Total Dysport®: Subjects received up to 3 doses of Dysport® 500 U/vial, 2 mL dilution on Day 1 of up to 3 treatment cycles. Subjects who were BoNT treatment naïve at the start of Study 169 received a starting dose of 500U/2 mL Dysport®, and subjects who were non-naïve to BoNT treatment received the same dose they had received on Day 1 of Study 169. Subjects received Dysport® by intramuscular injection into the same neck muscles that had been used for injection in Study 169. Retreatment occurred every 12 to 16 weeks, dependent on the investigator's clinical judgment. Follow-up visits occurred at Weeks 4 and 12 of each treatment cycle. Subjects were determined to have completed the study at Week 12 of Treatment Cycle 3. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-haemagglutinin complex (abobotulinumtoxinA).
Arm/Group | Total Dysport®
Number analyzed (Participants) | 112
Age, Customized [Number; unit: Participants]
  18-24 years | 0
  25-34 years | 1
  35-44 years | 13
  45-54 years | 34
  55-64 years | 33
  65-74 years | 26
  +75 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: TWSTRS Total Score at Week 4 and Week 12 for Treatment Cycles 1, 2 and 3.
Description: Mean TWSTRS total scores for Week 4 and Week 12 of treatment cycles 1, 2 and 3 are presented. The mean differences in the TWSTRS total scores from treatment cycle baseline (defined as Day 1 in each cycle) at the Week 4 and Week 12 visits for Treatment Cycles 1, 2 and 3 are also presented. The TWSTRS is an assessment scale used to measure the impact of CD on subjects, and comprises 3 subscales: severity, disability and pain, each of which is scored independently. The total score from the 3 subscales gives the TWSTRS total score with a value from 0 to 85 (best to worst). The score was assessed by the investigator at baseline and at all post-treatment visits of each treatment cycle.
Time Frame: Week 4 and 12 of treatment cycles 1, 2 and 3 (12 - 16 weeks duration each)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total Dysport®: Subjects received up to 3 doses of Dysport® 500 U/vial, 2 mL dilution on Day 1 of up to 3 treatment cycles. Subjects who were BoNT treatment naïve at the start of Study 169 received a starting dose of 500 U/2 mL Dysport®, and subjects who were non-naïve to BoNT treatment received the same dose they had received on Day 1 of Study 169. Subjects received Dysport® by intramuscular injection into the same neck muscles that had been used for injection in Study 169. Retreatment occurred every 12 to 16 weeks, dependent on the investigator's clinical judgment. Follow-up visits occurred at Weeks 4 and 12 of each treatment cycle. Subjects were determined to have completed the study at Week 12 of Treatment Cycle 3. Dysport® contains the neurotoxin Clostridium botulinum type A toxin-haemagglutinin complex (abobotulinumtoxinA).
Arm/Group | Total Dysport®
Number analyzed (Participants) | 112
units on a scale
  Mean TWSTRS score at Cycle 1-Day 1 | 37.7 (13.58)
  Mean TWSTRS score at Cycle 1-Week 4: number analyzed (Participants) | 102
  Mean TWSTRS score at Cycle 1-Week 4 | 30.1 (13.16)
  Mean TWSTRS score at Cycle 1-Week 12/Cycle 2-Day 1: number analyzed (Participants) | 98
  Mean TWSTRS score at Cycle 1-Week 12/Cycle 2-Day 1 | 32.6 (11.96)
  Mean TWSTRS score at Cycle 2-Week 4: number analyzed (Participants) | 96
  Mean TWSTRS score at Cycle 2-Week 4 | 27.0 (12.07)
  Mean TWSTRS score at Cycle 2-Week 12/Cycle 3-Day 1: number analyzed (Participants) | 92
  Mean TWSTRS score at Cycle 2-Week 12/Cycle 3-Day 1 | 31.1 (12.51)
  Mean TWSTRS score at Cycle 3-Week 4: number analyzed (Participants) | 91
  Mean TWSTRS score at Cycle 3-Week 4 | 27.4 (13.10)
  Mean TWSTRS score at Cycle 3-Week 12: number analyzed (Participants) | 92
  Mean TWSTRS score at Cycle 3-Week 12 | 30.1 (12.76)
Statistical Analysis 1: Comparison: Total Dysport®; Cycle 1-Day 1 vs Cycle 1-Week 4. The mean difference in the TWSTRS total scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 1 is presented; Test type: Superiority or Other; Mean Difference (Net) = -8.0, 95% CI 2-sided [-9.79 to -6.28], Standard Deviation 8.94
Statistical Analysis 2: Comparison: Total Dysport®; Cycle 1-Day 1 vs Cycle 1-Week 12. The mean difference in the TWSTRS total scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 1 is presented; Test type: Superiority or Other; Mean Difference (Net) = -5.0, 95% CI 2-sided [-7.36 to -2.68], Standard Deviation 11.68
Statistical Analysis 3: Comparison: Total Dysport®; Cycle 2-Day 1 vs Cycle 2-Week 4. The mean difference in the TWSTRS total scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 2 is presented; Test type: Superiority or Other; Mean Difference (Net) = -5.9, 95% CI 2-sided [-7.42 to -4.47], Standard Deviation 7.29
Statistical Analysis 4: Comparison: Total Dysport®; Cycle 2-Day 1 vs Cycle 2-Week 12. The mean difference in the TWSTRS total scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 2 is presented; Test type: Superiority or Other; Mean Difference (Net) = -1.8, 95% CI 2-sided [-3.37 to -0.27], Standard Deviation 7.49
Statistical Analysis 5: Comparison: Total Dysport®; Cycle 3-Day 1 vs Cycle 3-Week 4. The mean difference in the TWSTRS total scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 3 was determined; Test type: Superiority or Other; Mean Difference (Net) = -4.1, 95% CI 2-sided [-5.99 to -2.20], Standard Deviation 9.03
Statistical Analysis 6: Comparison: Total Dysport®; Cycle 3-Day 1 vs Cycle 3-Week 12. The mean difference in the TWSTRS total scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 3 was determined; Test type: Superiority or Other; Mean Difference (Net) = -1.1, 95% CI 2-sided [-3.11 to 0.81], Standard Deviation 9.42

2. Secondary Outcome: TWSTRS Total Scores at Pretreatment Baseline, Week 4 and Week 12 for Treatment Cycles 1, 2 and 3.
Description: The pretreatment baseline scores were defined as the TWSTRS measurement before Dysport® treatment in Study 169 for subjects who had received Dysport® in Study 169 and Day 1 of Study 170 for those subjects who had received placebo. Mean TWSTRS total scores for pretreatment baseline and for Week 4 and Week 12 of treatment cycles 1, 2 and 3 are presented. The mean differences in the TWSTRS total scores from pretreatment baseline scores at Week 4 and Week 12 of each treatment cycle are also presented. The TWSTRS is an assessment scale used to measure the impact of CD on subjects, and comprises 3 subscales: severity, disability and pain, each of which is scored independently. The total score from the 3 subscales gives the TWSTRS total score with a value from 0 to 85 (best to worst). The score was assessed by the investigator prior to study treatment at baseline for Studies 169 and 170 and at all post-treatment visits of each treatment cycle.
Time Frame: Week 4 and 12 of treatment cycles 1, 2 and 3 (12 - 16 weeks duration each)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 112
units on a scale
  Mean TWSTRS score at baseline for Study 169 | 42.2 (10.30)
  Mean TWSTRS score at Cycle 1-Week 4: number analyzed (Participants) | 102
  Mean TWSTRS score at Cycle 1-Week 4 | 30.1 (13.16)
  Mean TWSTRS score at Cycle 1-Week 12: number analyzed (Participants) | 98
  Mean TWSTRS score at Cycle 1-Week 12 | 32.6 (11.96)
  Mean TWSTRS score at Cycle 2-Week 4: number analyzed (Participants) | 96
  Mean TWSTRS score at Cycle 2-Week 4 | 27.0 (12.07)
  Mean TWSTRS score at Cycle 2-Week 12: number analyzed (Participants) | 92
  Mean TWSTRS score at Cycle 2-Week 12 | 31.1 (12.51)
  Mean TWSTRS score at Cycle 3-Week 4: number analyzed (Participants) | 91
  Mean TWSTRS score at Cycle 3-Week 4 | 27.4 (13.10)
  Mean TWSTRS score at Cycle 3-Week 12: number analyzed (Participants) | 92
  Mean TWSTRS score at Cycle 3-Week 12 | 30.1 (12.76)
Statistical Analysis 1: Comparison: Total Dysport®; Pretreatment baseline vs Cycle 1-Week 4. The mean difference in the TWSTRS total scores from baseline (pretreatment measurement before receiving Dysport® in Study 169 or for subjects who received placebo in Study 169, baseline was Day 1 of Cycle 1 of Study 170) at the Week 4 visit for Treatment Cycle 1 is presented; Test type: Superiority or Other; Mean Difference (Net) = -11.5, 95% CI 2-sided [-13.38 to -9.56], Standard Deviation 9.74
Statistical Analysis 2: Comparison: Total Dysport®; Pretreatment baseline vs Cycle 1-Week 12. The mean difference in the TWSTRS total scores from baseline (pretreatment measurement before receiving Dysport® in Study 169 or for subjects who received placebo in Study 169, baseline was Day 1 of Cycle 1 of Study 170) at the Week 12 visit for treatment Cycle 1 is presented; Test type: Superiority or Other; Mean Difference (Net) = -8.9, 95% CI 2-sided [-11.08 to -6.71], Standard Deviation 10.89
Statistical Analysis 3: Comparison: Total Dysport®; Pretreatment baseline vs Cycle 2-Week 4. The mean difference in the TWSTRS total scores from baseline (pretreatment measurement before receiving Dysport® in Study 169 or for subjects who received placebo in Study 169, baseline was Day 1 of Cycle 1 of Study 170) at the Week 4 visit for Treatment Cycle 2 is presented; Test type: Superiority or Other; Mean Difference (Net) = -14.4, 95% CI 2-sided [-16.74 to -12.11], Standard Deviation 11.43
Statistical Analysis 4: Comparison: Total Dysport®; Pretreatment baseline vs Cycle 2-Week 12. The mean difference in the TWSTRS total scores from baseline (pretreatment measurement before receiving Dysport® in Study 169 or for subjects who received placebo in Study 169, baseline was Day 1 of Cycle 1 of Study 170) at the Week 12 visit for Treatment Cycle 2 is presented; Test type: Superiority or Other; Mean Difference (Net) = -10.6, 95% CI 2-sided [-12.92 to -8.22], Standard Deviation 11.33
Statistical Analysis 5: Comparison: Total Dysport®; Pretreatment baseline vs Cycle 3-Week 4. The mean difference in the TWSTRS total scores from baseline (pretreatment measurement before receiving Dysport® in Study 169 or for subjects who received placebo in Study 169, baseline was Day 1 of Cycle 1 of Study 170) at the Week 4 visit for Treatment Cycle 3 is presented; Test type: Superiority or Other; Mean Difference (Net) = -14.6, 95% CI 2-sided [-17.18 to -12.10], Standard Deviation 12.19
Statistical Analysis 6: Comparison: Total Dysport®; Pretreatment baseline vs Cycle 3-Week 12. The mean difference in the TWSTRS total scores from baseline (pretreatment measurement before receiving Dysport® in Study 169 or for subjects who received placebo in Study 169, baseline was Day 1 of Cycle 1 of Study 170) at the Week 12 visit for Treatment Cycle 3 is presented; Test type: Superiority or Other; Mean Difference (Net) = -11.7, 95% CI 2-sided [-14.02 to -9.39], Standard Deviation 11.17

3. Secondary Outcome: Treatment Response in Treatment Cycle 3 Week 4.
Description: Treatment response was defined as a reduction in the TWSTRS total score of at least 30% from pretreatment baseline to the Week 4 visit in Treatment Cycle 3. The pretreatment baseline scores were defined as the TWSTRS measurement before Dysport® treatment in Study 169 for subjects who had previously received Dysport® in Study 169 and Day 1 of Study 170 for those subjects who had previously received placebo. The TWSTRS is an assessment scale used to measure the impact of CD on subjects, and comprises 3 subscales: severity, disability and pain, each of which is scored independently. The total score from the 3 subscales gives the TWSTRS total score with a value from 0 to 85 (best to worst). The score was assessed by the investigator prior to study treatment at baseline for Studies 169 and 170 and at all post-treatment visits of each treatment cycle. The proportion (percentage) of subjects who were treatment responders at Week 4 of Treatment Cycle 3 are presented.
Time Frame: Week 4 Treatment Cycle 3
Population: The safety population included all subjects who received at least 1 dose of study treatment, regardless of the amount of study treatment administered, and who had at least 1 safety record post-treatment or attended a post-treatment visit. For Treatment Cycle 3 there were 91 evaluable subjects.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Total Dysport®
Number analyzed (Participants) | 91
percentage of participants | 51.6 [40.93 to 62.26]

4. Secondary Outcome: TWSTRS Severity Subscale Score at Week 4 and Week 12 for Treatment Cycles 1, 2 and 3.
Description: Mean TWSTRS severity subscale scores for Week 4 and Week 12 of treatment cycles 1, 2 and 3 are presented. The mean differences in the TWSTRS severity subscale scores from treatment cycle baseline (defined as Day 1 in each cycle) at the Week 4 and Week 12 visits for treatment cycles 1, 2 and 3 are also presented. The TWSTRS is an assessment scale used to measure the impact of CD on subjects, and comprises 3 subscales: severity, disability and pain, each of which is scored independently. The total score from the 3 subscales gives the TWSTRS total score with a value from 0 to 85 (best to worst). The severity subscale gives a score from 0 to 35, with higher values indicating a worse outcome of physical findings of CD. The score was assessed by the investigator at baseline and at all post-treatment visits of each treatment cycle.
Time Frame: Weeks 4 and 12 of treatment cycle 1, 2 and 3 (12 - 16 weeks duration each)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 112
units on a scale
  Mean severity score at Cycle 1-Day 1 | 17.3 (4.69)
  Mean severity score at Cycle 1-Week 4: number analyzed (Participants) | 102
  Mean severity score at Cycle 1-Week 4 | 13.9 (5.21)
  Mean severity score Cycle 1-Week 12/Cycle 2-Day 1: number analyzed (Participants) | 98
  Mean severity score Cycle 1-Week 12/Cycle 2-Day 1 | 15.7 (4.97)
  Mean severity score at Cycle 2-Week 4: number analyzed (Participants) | 96
  Mean severity score at Cycle 2-Week 4 | 12.8 (4.97)
  Mean severity score Cycle 2-Week12/Cycle 3-Day 1: number analyzed (Participants) | 92
  Mean severity score Cycle 2-Week12/Cycle 3-Day 1 | 15.3 (4.87)
  Mean severity score at Cycle 3-Week 4: number analyzed (Participants) | 91
  Mean severity score at Cycle 3-Week 4 | 12.7 (5.78)
  Mean severity score at Cycle 3-Week 12: number analyzed (Participants) | 92
  Mean severity score at Cycle 3-Week 12 | 14.3 (5.29)
Statistical Analysis 1: Comparison: Total Dysport®; Cycle 1-Day 1 vs Cycle 1-Week 4. The mean difference in the TWSTRS severity subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 1 was determined; Test type: Superiority or Other; Mean Difference (Net) = -3.5, 95% CI 2-sided [-4.46 to -2.52], Standard Deviation 4.95
Statistical Analysis 2: Comparison: Total Dysport®; Cycle 1-Day 1 vs Cycle 1-Week 12. The mean difference in the TWSTRS severity subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 1 was determined; Test type: Superiority or Other; Mean Difference (Net) = -1.8, 95% CI 2-sided [-2.81 to -0.70], Standard Deviation 5.24
Statistical Analysis 3: Comparison: Total Dysport®; Cycle 2-Day 1 vs Cycle 2-Week 4. The mean difference in the TWSTRS severity subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 2 was determined; Test type: Superiority or Other; Mean Difference (Net) = -3.0, 95% CI 2-sided [-3.75 to -2.23], Standard Deviation 3.77
Statistical Analysis 4: Comparison: Total Dysport®; Cycle 2-Day 1 vs Cycle 2-Week 12. The mean difference in the TWSTRS severity subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 2 was determined; Test type: Superiority or Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.33 to 0.27], Standard Deviation 3.86
Statistical Analysis 5: Comparison: Total Dysport®; Cycle 3-Day 1 vs Cycle 3-Week 4. The mean difference in the TWSTRS severity subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 3 was determined; Test type: Superiority or Other; Mean Difference (Net) = -2.7, 95% CI 2-sided [-3.64 to -1.83], Standard Deviation 4.32
Statistical Analysis 6: Comparison: Total Dysport®; Cycle 3-Day 1 vs Cycle 3-Week 12. The mean difference in the TWSTRS severity subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 3 was determined; Test type: Superiority or Other; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.00 to -0.02], Standard Deviation 4.77

5. Secondary Outcome: TWSTRS Disability Subscale Score at Week 4 and Week 12 for Treatment Cycles 1, 2 and 3.
Description: Mean TWSTRS disability subscale scores for Week 4 and Week 12 of treatment cycles 1, 2 and 3 are presented. The mean difference in the TWSTRS disability subscale scores from treatment cycle baseline (defined as Day 1 in each cycle) at the Week 4 and Week 12 visits for Treatment Cycles 1, 2 and 3 are also presented. The TWSTRS is an assessment scale used to measure the impact of CD on subjects, and comprises 3 subscales: severity, disability and pain, each of which is scored independently. The total score from the 3 subscales gives the TWSTRS total score with a value from 0 to 85 (best to worst). The disability subscale is a 6-item scale and each item is rated on a 6-point scale with higher values indicating the highest degree of disability. The score was assessed by the investigator at baseline and at all post-treatment visits of each treatment cycle.
Time Frame: Weeks 4 and 12 of treatment cycle 1, 2 and 3 (12 - 16 weeks duration each)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 112
units on a scale
  Mean disability score at Cycle 1-Day 1 | 11.5 (6.63)
  Mean disability score at Cycle1-Week 4: number analyzed (Participants) | 102
  Mean disability score at Cycle1-Week 4 | 8.8 (6.41)
  Mean disability score Cycle1-Week 12/Cycle 2-Day 1: number analyzed (Participants) | 98
  Mean disability score Cycle1-Week 12/Cycle 2-Day 1 | 9.4 (5.64)
  Mean disability score at Cycle 2-Week 4: number analyzed (Participants) | 96
  Mean disability score at Cycle 2-Week 4 | 7.9 (5.76)
  Mean disability score Cycle2-Week 12/Cycle 3-Day 1: number analyzed (Participants) | 92
  Mean disability score Cycle2-Week 12/Cycle 3-Day 1 | 8.7 (5.82)
  Mean disability score at Cycle 3-Week 4: number analyzed (Participants) | 91
  Mean disability score at Cycle 3-Week 4 | 8.1 (6.07)
  Mean disability score at Cycle 3-Week 12: number analyzed (Participants) | 92
  Mean disability score at Cycle 3-Week 12 | 8.6 (6.41)
Statistical Analysis 1: Comparison: Total Dysport®; Cycle 1-Day 1 vs Cycle 1-Week 4. The mean difference in the TWSTRS disability subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 1 was determined; Test type: Superiority or Other; Mean Difference (Net) = -2.9, 95% CI 2-sided [-3.64 to -2.12], Standard Deviation 3.86
Statistical Analysis 2: Comparison: Total Dysport®; Cycle 1-Day 1 vs Cycle 1-Week 12.The mean difference in the TWSTRS disability subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 1 was determined; Test type: Superiority or Other; Mean Difference (Net) = -1.8, 95% CI 2-sided [-2.79 to -0.86], Standard Deviation 4.82
Statistical Analysis 3: Comparison: Total Dysport®; Cycle 2-Day 1 vs Cycle 2-Week 4. The mean difference in the TWSTRS disability subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 2 was determined; Test type: Superiority or Other; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.44 to -1.04], Standard Deviation 3.47
Statistical Analysis 4: Comparison: Total Dysport®; Cycle 2-Day 1 vs Cycle 2-Week 12. The mean difference in the TWSTRS disability subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 2 was determined; Test type: Superiority or Other; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.55 to -0.12], Standard Deviation 3.46
Statistical Analysis 5: Comparison: Total Dysport®; Cycle 3-Day 1 vs Cycle 3-Week 4. The mean difference in the TWSTRS disability subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 3 was determined; Test type: Superiority or Other; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.45 to 0.12], Standard Deviation 3.75
Statistical Analysis 6: Comparison: Total Dysport®; Cycle 3-Day 1 vs Cycle 3-Week 12.The mean difference in the TWSTRS disability subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 3 was determined; Test type: Superiority or Other; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.85 to 0.70], Standard Deviation 3.73

6. Secondary Outcome: TWSTRS Pain Subscale Score at Week 4 and Week 12 for Treatment Cycles 1, 2 and 3.
Description: Mean TWSTRS pain subscale scores for Week 4 and Week 12 of treatment cycles 1, 2 and 3 are presented. The mean difference in the TWSTRS pain subscale scores from treatment cycle baseline (defined as Day 1 in each cycle) at the Week 4 and Week 12 visits for Treatment Cycles 1, 2 and 3 are also presented. The TWSTRS is an assessment scale used to measure the impact of CD on subjects, and comprises 3 subscales: severity, disability and pain, each of which is scored independently. The total score from the 3 subscales gives the TWSTRS total score with a value from 0 to 85 (best to worst). The pain subscale gives a score from 0 to 20, with higher values indicating greater pain experienced. The score was assessed by the investigator at baseline and at all post-treatment visits of each treatment cycle.
Time Frame: Week 4 and 12 of treatment cycles 1, 2 and 3 (12 - 16 weeks duration each)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Dysport®
Number analyzed (Participants) | 112
units on a scale
  Mean pain score at Cycle 1-Day 1 | 9.0 (5.32)
  Mean pain score at Cycle 1-Week 4: number analyzed (Participants) | 102
  Mean pain score at Cycle 1-Week 4 | 7.4 (5.10)
  Mean pain score at Cycle 1-Week 12/Cycle 2-Day 1: number analyzed (Participants) | 98
  Mean pain score at Cycle 1-Week 12/Cycle 2-Day 1 | 7.5 (5.03)
  Mean pain score at Cycle 2- Week 4: number analyzed (Participants) | 96
  Mean pain score at Cycle 2- Week 4 | 6.3 (5.11)
  Mean pain score at Cycle 2-Week 12/Cycle 3-Day 1: number analyzed (Participants) | 92
  Mean pain score at Cycle 2-Week 12/Cycle 3-Day 1 | 7.2 (4.98)
  Mean pain score at Cycle 3-Week 4: number analyzed (Participants) | 91
  Mean pain score at Cycle 3-Week 4 | 6.5 (5.01)
  Mean pain score at Cycle 3-Week 12: number analyzed (Participants) | 92
  Mean pain score at Cycle 3-Week 12 | 7.1 (4.85)
Statistical Analysis 1: Comparison: Total Dysport®; Cycle 1-Day 1 vs Cycle 1-Week 4. The mean difference in the TWSTRS pain subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 1 was determined; Test type: Superiority or Other; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.39 to -0.92], Standard Deviation 3.74
Statistical Analysis 2: Comparison: Total Dysport®; Cycle 1-Day 1 vs Cycle 1-Week 12. The mean difference in the TWSTRS pain subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 1 was determined; Test type: Superiority or Other; Mean Difference (Net) = -1.4, 95% CI 2-sided [-2.22 to -0.66], Standard Deviation 3.88
Statistical Analysis 3: Comparison: Total Dysport®; Cycle 2-Day 1 vs Cycle 2-Week 4.The mean difference in the TWSTRS pain subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 2 was determined; Test type: Superiority or Other; Mean Difference (Net) = -1.2, 95% CI 2-sided [-1.84 to -0.58], Standard Deviation 3.12
Statistical Analysis 4: Comparison: Total Dysport®; Cycle 2-Day 1 vs Cycle 2-Week 12. The mean difference in the TWSTRS pain subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 2 was determined; Test type: Superiority or Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.08 to 0.18], Standard Deviation 3.04
Statistical Analysis 5: Comparison: Total Dysport®; Cycle 3-Day 1 vs Cycle 3-Week 4. The mean difference in the TWSTRS pain subscale scores from treatment cycle baseline (Day 1) at the Week 4 visit for Treatment Cycle 3 was determined; Test type: Superiority or Other; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.57 to 0.19], Standard Deviation 4.20
Statistical Analysis 6: Comparison: Total Dysport®; Cycle 3-Day 1 vs Cycle 3-Week 12. The mean difference in the TWSTRS pain subscale scores from treatment cycle baseline (Day 1) at the Week 12 visit for Treatment Cycle 3 was determined; Test type: Superiority or Other; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.85 to 0.73], Standard Deviation 3.78

ADVERSE EVENTS:
Time Frame: In Study 170 AEs were collected from Day 1 of Treatment Cycle 1 up to the end of study (Week 12 of Treatment Cycle 3)/early withdrawal. For subjects who received Dysport® in Study 169, AEs were collected over 4 Dysport® dosing cycles; 1 Dysport® dosing cycle from Study 169 and 3 Dysport® dosing cycles from Study 170 (period of up to 49 weeks). For subjects who received placebo in Study 169, AEs were collected in 3 Dysport® dosing cycles from Study 170 (period of up to 36 weeks).
Description: Serious and non-serious treatment emergent AEs are presented for all Dysport® dosing cycles in Study 169 and Study 170. The safety population consisted of all randomised subjects who received at least 1 dose of study treatment regardless of the amount of study treatment administered and who had at least 1 safety record post-treatment or attended a post-treatment visit.
Arm/Group | Total Dysport®
Serious Adverse Events (participants affected / at risk) | 7/112
Other Adverse Events (participants affected / at risk) | 70/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Dysport® (N=112)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Dysport® (N=112)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 12 (16)
Neck Pain (Musculoskeletal and connective tissue disorders) | 12 (13)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myofascial Pain Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Sensation of Heaviness (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal Deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (7)
Dizziness (Nervous system disorders) | 3 (5)
Migraine (Nervous system disorders) | 3 (3)
Aphasia (Nervous system disorders) | 1 (1)
Balance Disorder (Nervous system disorders) | 1 (1)
Burning Sensation (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Head Discomfort (Nervous system disorders) | 1 (1)
Hyporeflexia (Nervous system disorders) | 1 (1)
Movement Disorder (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Tension Headache (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 12 (15)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Dry Mouth (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Diverticulum Intestinal (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Candidiasis (Infections and infestations) | 1 (1)
Ear Infection (Infections and infestations) | 1 (1)
Gastrointestinal Viral Infection (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Ligament Injury (Injury, poisoning and procedural complications) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1)
Tooth Injury (Injury, poisoning and procedural complications) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Injection Site Pain (General disorders) | 1 (1)
Injection Site Reaction (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vision Blurred (Eye disorders) | 4 (4)
Dry Eye (Eye disorders) | 1 (1)
Eye Pain (Eye disorders) | 1 (1)
Ocular Hyperaemia (Eye disorders) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 1 (1)
Barium Swallow (Investigations) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1)
Blood Cholesterol Increased (Investigations) | 1 (1)
Blood Testosterone Decreased (Investigations) | 1 (1)
Blood Triglycerides Increased (Investigations) | 1 (2)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Sleep Disorder (Psychiatric disorders) | 1 (1)
Tic (Psychiatric disorders) | 1 (1)
Breast Mass (Reproductive system and breast disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Pelvic Fluid Collection (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 1 (2)
Motion Sickness (Ear and labyrinth disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Endodontic Procedure (Surgical and medical procedures) | 1 (1)
Rotator Cuff Repair (Surgical and medical procedures) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No